CLINICAL TRIAL: NCT04576715
Title: Promoting Recovery in Children Who Sustain a Mild Traumatic Brain Injury: mTBI Evaluation and Management (TEaM)
Brief Title: TBI Evaluation and Management (TEaM)
Acronym: TEaM
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Emory University (Other)
Collaborators: Children's Healthcare of Atlanta (Other)
Responsible Party: Principal Investigator, David Wright, Professor, Emory University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IRB00108674
Record Dates: First submitted 2020-10-01; First posted 2020-10-06 (Actual); Last update posted 2025-02-25 (Actual); Status verified 2025-02

CONDITIONS: Mild Traumatic Brain Injury
Keywords: mTBI; Brain injury; Emergency medicine; Urgent care; Primary care; Concussion; Pediatrics
MeSH Terms: conditions — Brain Concussion; Brain Injuries | interventions — Standard of Care

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- TEaM Intervention Group (Experimental): Dedicated Provider Education plus Information Technology Support. The IT support includes addition of an eMR concussion screening, followed by an alert to the provider, followed by a structured assessment / evaluation template.
  Interventions: Behavioral: TEaM Intervention
- Control Group (Active Comparator): Standard medical protocol for the management of mTBI in children. This group will not receive interventional Provider Training on the TEaM concussion evaluation examination and utilization of the eMR template.
  Interventions: Behavioral: Standard of Care

INTERVENTIONS:
Behavioral: TEaM Intervention — Multi-setting mTBI (mild traumatic brain injury) Evaluation and Management Intervention incorporates provider education and information technology support systems, based on the best available evidence and tailored to a specific environment (acute care setting vs primary care clinic). Facilitates linkages between providers (ED/UC to primary care) and systems (healthcare to school).
  * Provider Training Modules: Training includes decision-making support alerted by positive triage screening and concussion-specific eMR template
  * Management based on current best practices (however, may have additional education from the provider training)
  * Return to school letters
  * Primary Care Follow Up
  Other Names: TEaM
  Arms: TEaM Intervention Group
Behavioral: Standard of Care — Continue with CHOA current best practices for mTBI:
  * No TEaM Provider training (but will be offered to all providers at end of study)
  * Will not be trained on utilization and implementation of the concussion screening alert and eMR template
  Arms: Control Group

SUMMARY:
The purpose of this study is to evaluate a multi-disciplinary, multi-setting intervention with the goal of improving outcomes for children who have experienced a mild traumatic brain injury (mTBI). The project aims to improve and support mTBI diagnosis and management, and improve critical decision making by clinicians during their interaction with the injured child, their family, and their school.

DETAILED DESCRIPTION:
Emergency, urgent care, and primary care providers participating in the study will be block randomized in a 1:1 ratio by practice type to receive the intervention or continue with their standard practice. All enrolled clinicians (both trained and control providers) patients they care for will be screened for inclusion in the trial.

Additionally, a pre/post intervention will be layered upon the randomized educational intervention to evaluate the effects of the information technology decision support tool (i.e. eMR) in isolation of the clinician education intervention. The 32-month mTBI patient enrollment period will be divided into two 16 months segments. The first 16 months will be without the eMR intervention being visible, and the remaining 16 months post eMR screening and decision support deployment in the ED and UC. This study design allows us to evaluate the independent and interactive effects of the decision support tool and educational intervention.

Enrolled children will be followed for up to three months post injury to ascertain the effect of the interventions on the primary aim (reduction of school problems/performance) and secondary aims.

ELIGIBILITY:
PROVIDER INCLUSION CRITERIA

* Actively practicing physician or APP in the CHOA System
* Primary practice in either ED, UC, and/or PCP

PROVIDER EXCLUSION CRITERIA

* Inability or unwillingness to provide written/electronic informed consent
* Unable to fulfill study training / education requirements

CHILD INCLUSION CRITERIA - RETROSPECTIVE

* School age (5-18 yoa)
* Evaluated in ED / UC / PCP within 72 hours of injury
* Discharged home from ED / UC / PCP (e.g., not admitted to hospital)

CHILD EXCLUSION CRITERIA - RETROSPECTIVE

* Non-English speaking
* Known severe developmental delay or known severe psychiatric history
* Known prior severe brain injury
* Known mTBI within past 3 months
* First mTBI visit outside of CHOA network

CHILD INCLUSION CRITERIA - PROSPECTIVE

* Meets above inclusion for retrospective portion plus:
* mTBI likely present as defined by:
* Positive diagnosis by clinician or mTBI OR
* Positive triage screen plus positive symptom checklist

CHILD EXCLUSION CRITERIA - PROSPECTIVE

* Does not meet above exclusion for retrospective portion plus:
* Requests to Opt-Out via e-mail or first phone contact
* Inability or unwillingness to provide verbal informed telephone consent/assent

Min Age: 5 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 1000 (Estimated)
Dates: Start 2022-08-19 (Actual); Primary Completion 2026-06 (Estimated); Study Completion 2027-01 (Estimated)

PRIMARY OUTCOMES:
Change in CLASS survey score | 1 week, 2 week and 1 month post return to school
  Concussion Learning Assessment and School Survey (CLASS), identifies the types of problems students experienced across all grades. Total score range 0-42 (14 individual items rated 0-3, 0 = no problem, 3 = significant problem). Higher score reflects a greater problem/ worse outcome.
Change in Post-concussion symptom inventory (PCSI) total score | 1 week, 2 week and 1 month post return to school
  Change in Post-concussion symptom inventory (PCSI). Total score range, 0-24 (4 symptoms on a 0-6 scaling). Higher score reflects a greater problem/worse outcome.
Change in Peds-QL score | 1 week, 2 week and 1 month post return to school
  Pediatric Quality of Life (PedsQL) scale, includes 23 items, rated 0-4 (assesses different areas of function (physical, emotional, social, school) to determine if the child is having any problems with various tasks in each functional area and if so, how often the difficulty occurs).
  4 sub scales (general health 8 items 0-4 scaling, 0-32 total; social 5 items, 0-4 scaling, 0-20; school 5 items, 0-4 scaling, 0-20; emotional 5 items, 0-4 scaling, 0-20, 0=it is never a problem, 4= it is almost always a problem). Higher raw score reflects worse overall quality of life. Items are calculated and transformed into an overall score with a range of 0-to-100 points, with 100 points indicating better HRQoL.
Post-concussion symptom inventory (PCSI) total score at 3 months post injury | 3 months post injury
  Persistent post-mTBI symptoms as measured by the PCSI total score at 3 months post injury.
  Total score range, 0-24 (4 symptoms on a 0-6 scaling). Higher score reflects a greater problem/worse outcome.
Time to return to full activity post injury | Up to 3 months post-intervention
  Measured by serial PCSI and return to activity. PCSI Total score (PPCS-Persistent Post-Concussive Symptoms - will be calculated via the PCSI Total Score with scores classified as "Recovered" or "Non-Recovered (PPCS)" based on the Reliable Change Metrics that reflect recovery or not (e.g., for Parent and Adolescent PCSI Total RAPID score <5 indicates symptom recovery). Total score ranges from 0 to 100%. Lower % with PPCS in Intervention group compared to Control indicates better study outcome.

SECONDARY OUTCOMES:
Primary Care Physician (PCP) follow up visits | 3 months post-intervention
  Number of PCP visits for concussion during 3 month follow-up period.
Number of letters sent to school | 2 weeks post-injury
  Number of Primary care Physician (PCP) letters sent to school within 2 weeks post-injury

CONTACTS AND LOCATIONS:
Overall Officials: David Wright, MD, Principal Investigator — Emory University
Locations (3):
- United States (3):
  - Children's Healthcare of Atlanta (CHOA) - Egleston Emergency Department, Atlanta, Georgia
  - Children's Healthcare of Atlanta- Forsyth, Northpoint and Town Center Urgent Care Centers, Atlanta, Georgia
  - Children's Healthcare of Atlanta- Primary Care Offices, Atlanta, Georgia

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol, SAP
Time Frame: A year after study closure. No end date
Access Criteria: Data will be publicly available via the internet in a way that the CDC/CIO dictate, through a CDC data repository, at which point the PIs will no longer have stewardship over the data.